CLINICAL TRIAL: NCT06438185
Title: Evaluation of The Efficacy And Safety of An Irreversible Electroporation (IRE) System For Treatment of Inferior Turbinate Hypertrophy With Nasal Obstruction
Brief Title: Efficacy And Safety of An IRE System For Treatment of Inferior Turbinate Hypertrophy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ENTire Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 0157
Record Dates: First submitted 2024-05-23; First posted 2024-05-31 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Inferior Turbinate Hypertrophy; Nasal Obstruction; Turbinate; Hypertrophy Mucous Membrane
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Intervention Model Description: Irreversible Electroporation (IRE) System for Inferior Turbinate Hypertrophy with Nasal Obstruction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enlarged Inferior Turbinate(s) will be reduced by ENTire IRE System. (Experimental): The bi-polar IRE System locally applies short, high-voltage (HV) pulses, increasing the permeability of tissue cells, creating non-thermal irreversible electroporation (NTIRE). The energy is transferred via bipolar forceps and causes irreversible cell membrane perforation and apoptosis. This results in tissue reduction within 2-4 weeks after treatment.
  Interventions: Device: IRE System

INTERVENTIONS:
Device: IRE System — Irreversible Electroporation (IRE) System for Inferior Turbinate Hypertrophy with Nasal Obstruction.
  Other Names: ENtire IRE System

SUMMARY:
The purpose of the IRE System is to address the clinical need for reducing the volume of hypertrophic inferior turbinate(s) causing nasal obstruction while minimizing side effects and complications. Procedure time will also be reduced. The IRE System is designed to be more comfortable for patients, as it employs a noninvasive procedure using a high voltage pulsed electric field to create irreversible nanopores in the cell membrane, leading to cell death and the reduction of the inferior turbinate volume.

DETAILED DESCRIPTION:
The purpose of the IRE System is to address the clinical need for reducing the volume of hypertrophic inferior turbinate(s) causing nasal obstruction while minimizing side effects and complications. Procedure time will also be reduced. The IRE System is designed to be more comfortable for patients, as it employs a noninvasive procedure using a high voltage pulsed electric field to create irreversible nanopores in the cell membrane, leading to cell death and the reduction of tonsil volume. On basis of these finding and in view of the known safety profile (refer to Chen et.al ) and efficacy of current technologies, the purpose of the current study is to prospectively determine the efficacy and safety of the IRE System in interior turbinate reduction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70 years.
* Nasal Obstruction Symptom Evaluation (NOSE) score of ≥ 60 at the Baseline.
* Hypertrophy of the inferior turbinate is the primary cause of the patient's nasal obstruction based on vasoconstriction test.
* Did not improve with medical treatment, including topical nasal steroids for nasal obstruction for at least three months.

Exclusion Criteria:

* Age below 18 years
* Patients with a pacemaker or similar electro stimulator
* Patients with caudal septal deviation that narrows the anterior nasal valve.
* Patients with nasal polyps/tumors.
* Patients with chronic rhinosinusitis.
* Patients with Eosinophilia
* Patients for whom the anesthesia involves high risk.
* Patients with Epilepsy or other condition involving convulsions.
* Patients with an inability to give informed consent and to complete self-reported questionnaires.
* Patients with an inability to cooperate for treatment and follow-up.
* Patients with severe heart disease.
* Pregnancy or breastfeeding.
* Previous inferior turbinate surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in Nasal Obstruction Symptom Evaluation Scale (NOSE) | 3 months post treatment
  A change of > 20% in Nasal Obstruction Symptom Evaluation Scale scale and a > 20% in the Nasal Obstruction VAS score as compared to screening visit.

SECONDARY OUTCOMES:
A Sinonasal Outcome Test (SNOT-22) score | 3 months post treatment
  A Sinonasal Outcome Test (SNOT-22) score improvement by at least a 8.9 point reduction at 3 months post treatment.
Pain Visual Analog Scale (VAS) | up to 1 week post treatment and through study subject completion
  Low to moderate Pain VAS (VAS/Pain VAS) score (1-3 on a VAS Scale) post treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Saint Mary Hospital, Bucharest, Romania
- Republican Specialized Scientific and Practical Medical Center for Otorhinolaryngology and Head and Neck Diseases, Tashkent, Yashnabad District, Uzbekistan

IPD SHARING:
Plan to Share IPD: No